CLINICAL TRIAL: NCT06324396
Title: IMProving DRug Dosing and Outcomes for Single VEntricle Patients With Fontan Associated Liver Disease
Acronym: IMPROVE-FALD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jon Wagner, Director, Division of Clinical Pharmacology, Toxicology, and Therapeutic Innovation, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002974; 5T32HD069038 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-03-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Fontan Circulation
Keywords: Fontan; FALD
MeSH Terms: interventions — Sildenafil Citrate; Tablets; Pravastatin; Glycation End Products, Advanced

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, prospective, investigation to quantify the effects of liver congestion and fibrosis has on hepatic statin transport (SA1) and response (SA2) in children, adolescents, and young adults with Fontan circulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment Arm (Experimental): Assessment group will receive a single dose of oral sildenafil and oral pravastatin.
  Interventions: Drug: Sildenafil 10mg oral tablet (participants <20kg), or 20mg oral tablet (participants ≥20kg); Drug: Pravastatin 20 mg oral tablet (ages <13 years), or 40 mg oral tablet (≥14 years)

INTERVENTIONS:
Drug: Sildenafil 10mg oral tablet (participants <20kg), or 20mg oral tablet (participants ≥20kg) — A single oral dose of sildenafil will be administered to all study subjects.
Drug: Pravastatin 20 mg oral tablet (ages <13 years), or 40 mg oral tablet (≥14 years) — A single oral dose of pravastatin will be administered to all study subjects.

SUMMARY:
This is a single center, open-label, prospective, investigation to quantify the effects liver congestion and fibrosis has on hepatic drug metabolism and transport in children, adolescents, and young adults with Fontan circulation.

ELIGIBILITY:
Inclusion Criteria:

* > 8 years
* Status Post Fontan Completion
* Ability to provide informed permission-assent (<18 years) or consent (≥18 years)
* Fasting overnight (~8 hours)

Exclusion Criteria:

* Pregnancy
* Non-fasting
* Non-removable metal in body or where magnetic resonance imaging (MRI) is considered unsafe
* Sildenafil and/or Pravastatin therapy within last 2 months
* History of underlying or laboratory evidence of underlying intestinal, metabolic, autoimmune, renal disease that can alter Sildenafil and Pravastatin disposition (absorption, metabolism, distribution, or clearance)
* Pharmacotherapy that interacts with Sildenafil (cytochrome P450 3A4 and P450 3A5 (CYP3A4/5) inducers/inhibitors) and/or Pravastatin (organic anion transporting polypeptide (OATP1B1) inducers/inhibitors)
* Inability to swallow a tablet
* >5X the age-specific upper limit of normal for aspartate aminotransferase (AST) and alanine aminotransferase (ALT), total and conjugated bilirubin
* Diarrhea in the last 24 hours *History of solid organ transplantation

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sildenafil concentration as measured by area under the curve (AUC) | 2 years
  Area under the time-exposure curve (AUC 0-n) for sildenafil as determinants of the dose-exposure relationship.
Pravastatin concentration as measured by area under the curve (AUC) | 2 years
  Area under the time-exposure curve (AUC 0-n) for pravastatin as determinants of the dose-exposure relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wagner, DO, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States